CLINICAL TRIAL: NCT07341568
Title: Leptin and Irisin Hormonal Crosstalk in Cognitive Health Among Aging Individuals: The Modulatory Role of Exercise
Brief Title: Exercise-Modulated Cognitive Hormones
Status: Completed | Type: Observational
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Sami Gabr, clinical Professor, King Saud University
Other Study IDs: RRC-2023-029
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Cognitive Impairment; Healthy Participants
Keywords: cognitive capacity, Leptin, Irisin, BDNF hormones
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood samples were obtained from all subjects at 0800 h after an overnight fast before and after the training program Venous blood samples (5 mL) were collected into plain tubes, the samples were allowed to clot for half an hour following which samples were centrifuged for 15 minutes at 2000 rpm. Samples were given a coded study identification number and were stored frozen at 80°C until analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- participants with cognitive impairment: subjects with cognitive imparment as measured by the Loewenstein Occupational Therapy Cognitive Assessment (LOTCA) battery.
- healthy goup: Subjects are healthy without any diseases and are normal as estimated by the Loewenstein Occupational Therapy Cognitive Assessment (LOTCA) battery.

SUMMARY:
Investigating the influence of a 12-week exercise regimen structured thrice weekly on cognitive capacity, and related hormones like Leptin, Irisin, BDNF hormones, antioxidant status, and inflammatory cytokines, whether these modulations potentially enhance neuroprotection and mitigate age-related cognitive impairment among healthy adults.

DETAILED DESCRIPTION:
To elucidate the potential role of exercise as a buffer of cognitive impairment among healthy adults. We thought to investigate the effect of supervised aerobic training of moderate intensity on related hormones like Leptin, Irisin, BDNF hormones, antioxidant status, and inflammatory cytokines, whether these modulations potentially enhance neuroprotection and mitigate age-related cognitive impairment among healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Sixty healthy individuals, aged 50 to 80 years (30 men/30 women), were invited to participate in this study after provided with informed consent and were included in this study. Also, all participants were of a sedentary lifestyle, with little or no physical activity during daily routine activities like work and transportation

Exclusion Criteria:

* To ensure accurate results, participants with obesity (BMI) ≥35 kg/m2.), physical impairments, movement limitations, chronic illnesses, such as kidney or liver diseases, or severe diabetes-related complications such as neuropathy, retinopathy, neuromuscular issues, cardiopulmonary conditions, or disorders affecting eating, the endocrine system, immune system, or mental health or those who undergoing glucocorticoid medication were excluded from this study

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sixty healthy individuals, aged 50 to 80 years (30 men/30 women), were invited to participate in this study after provided with informed consent.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2025-06-15 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Assessment of cognitive abilities | 6 months
  Trained research assistants assessed the cognitive abilities of older adult's pre and post supervised aerobic exercise using the Loewenstein Occupational Therapy Cognitive Assessment (LOTCA) battery. Assessments required between 45 and 90 minutes.
2- Leisure-time physical activity (LTPA) | 6 months
  A verified questionnaire was utilized to assess physical activity, specifically focusing on leisure-time physical activity (LTPA). In alignment with previous findings, we measured the weekly energy expenditure in terms of metabolic equivalents per hour per week (T-LPTA-MET/H/W
3-Assessment of apoptotic-related proteins | 6 month
  Blood serum samples were collected from all participants in the early hours after a night of fasting, both before and after the exercise training regimen, to analyze apoptosis-related proteins. Immunoassay methods were used to measure serum Bcl-2 and cytochrome c levels. This involved using ELISA kits specifically designed for Bcl-2 (Cat# QIA23, Oncogene Research Products, Germany) and cytochrome c (Zymed ELISA Kit, Cat. No. 99-0040). Furthermore, the quantification of p53 concentration in the serum was determined utilizing a single-step enzyme-immunoassay ELISA kit (Catalog Number 11 828 789 001; Roche Diagnostics GmbH, Roche Applied Science, Germany) based on photometric methods.

SECONDARY OUTCOMES:
biochemical analysis of hormones, antioxidant enzymes, before and after exercise training | 6 month
  The levels of Leptin, Irisin, BDNF hormones, antioxidant status, and inflammatory cytokines were identified from the serum of all subjects, healthy and cognitively impaired subjects, before and after exercise sessions

CONTACTS AND LOCATIONS:
Overall Officials: Sami Gabr, Principal Investigator — Medical Microbiology Dept, ImmunityUnit,Faculty of Medicine, Mansoura University, Egypt
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No